CLINICAL TRIAL: NCT04603495
Title: A Phase 3, Randomized, Double-blind, Active-Control Study of Pelabresib (CPI-0610) and Ruxolitinib vs. Placebo and Ruxolitinib in JAKi Treatment Naive MF Patients
Brief Title: Phase 3 Study of Pelabresib (CPI-0610) in Myelofibrosis (MF) (MANIFEST-2)
Acronym: MANIFEST-2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDAK539A12301; 2023-507954-34-00 (Registry Identifier: EU CT Number); CPI 0610-04 (Other: Constellation Pharmaceuticals)
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Results first posted 2024-10-28 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Myelofibrosis; Primary Myelofibrosis; Post-polycythemia Vera Myelofibrosis; Post-essential Thrombocythemia Myelofibrosis
Keywords: Pelabresib; Ruxolitinib
MeSH Terms: conditions — Primary Myelofibrosis | interventions — ruxolitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study has a double-blind design in which patients and investigators are blinded to study drug; study drugs will be packaged identically. All patients will be randomly assigned to either treatment group in a 1:1 ratio. The blind should only be broken in the case of emergency.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pelabresib + ruxolitinib (Experimental): Pelabresib monohydrate tablets + ruxolitinib phosphate tablets
  Interventions: Drug: Pelabresib; Drug: Ruxolitinib
- Placebo + ruxolitinib (Active Comparator): Matching placebo tablets + ruxolitinib phosphate tablets
  Interventions: Drug: Ruxolitinib; Drug: Placebo

INTERVENTIONS:
Drug: Pelabresib — Double-blind treatment (pelabresib or matching placebo) will be administered daily for 14 consecutive days followed by a 7-day break, which is considered 1 cycle of treatment (1 cycle = 21 days).
  Pelabresib is a small molecule inhibitor of BET proteins with a novel mechanism of action and potential for disease-modifying effects in MF.
  Arms: Pelabresib + ruxolitinib
Drug: Ruxolitinib — Ruxolitinib is a JAK inhibitor and a current, approved treatment option for MF.
Drug: Placebo — Placebo tablets are designed to match pelabresib tablets. Each placebo tablet contains no active pharmaceutical ingredient and is visibly identical to experimental drug in size, shape, and packaging. Placebo dosing follows the same dosing conventions as pelabresib.
  Arms: Placebo + ruxolitinib

SUMMARY:
A Phase 3, randomized, blinded study comparing pelabresib (CPI-0610) and ruxolitinib with placebo and ruxolitinib in myelofibrosis (MF) patients that have not been previously treated with Janus kinase inhibitors (JAKi). Pelabresib is a small molecule inhibitor of bromodomain and extra-terminal (BET) proteins.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Confirmed diagnosis of myelofibrosis (primary, post-polycythemia vera, or post essential thrombocythemia)
* Adequate hematologic, renal, and hepatic function
* Have at least 2 symptoms with an average score ≥ 3 or an average total score of ≥ 10 over the 7-day period prior to randomization using the MFSAF v4.0
* Prognostic risk-factor score of Intermediate-1 or higher per Dynamic International Prognostic Scoring System (DIPSS) scoring system
* Spleen volume of ≥ 450 cm^3
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2

Exclusion Criteria:

* Splenectomy or splenic irradiation in the previous 6 months
* Chronic or active conditions and/or concomitant medication use that would prohibit treatment
* Had prior treatment with any JAKi or BET inhibitor for treatment of a myeloproliferative neoplasm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2027-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (156):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Ironwood Physicians P.C. dba Ironwood Cancer and Research Centers, Chandler, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Mayo Clinic, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Decatur Memorial Hospital Cancer Care Center of Decatur/Cancer Care Specialists of IL, Decatur, Illinois
  - Franciscan Health/Indiana blood and Marrow Transplantation, Indianapolis, Indiana
  - Norton Cancer Institute, St. Matthews Campus, Louisville, Kentucky
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College- New York Presbyterian Hospital, New York, New York
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center - San Antonio, San Antonio, Texas
  - Center for Blood Disorders and Cellular Therapy, Swedish Cancer Institute, Seattle, Washington
- Australia (6):
  - Icon Cancer Centre, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Health, Clayton, Victoria
  - Peninsula Private Hospital Clinical Trials Unit, Frankston, Victoria
  - USC Clinical Trials Centre Sunshine Coast Haematology and Oncology Clinic, Buderim
  - One Clinical Research PTY LTD, Nedlands
- Austria (4):
  - LKH - Universitätsklinikum Graz; Abteilung für Hämatologie, Graz
  - Krankenhaus der Elisabethinen Linz, Linz
  - Kepler University Hospital, Linz
  - University Hospital Salzburg, Salzburg
- Belgium (5):
  - ZNA, Antwerp
  - Cliniques universitaires Saint-Luc, Brussels
  - Hôpital de Jolimont, La Louvière
  - UZ Leuven, Leuven
  - Domaine Universitaire du Sart Tilman, Liège
- Canada (5):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - London Health Sciences Center - Victoria Hospital, London, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- Czechia (2):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - University Hospital Olomouc, Olomouc
- France (9):
  - Amiens South Hospital univerisy - Hopital Sud, Amiens
  - Centre Hospitalier, Le Mans
  - Hôpital l'Archet 1, Nice
  - Gard Cancer Institute, Nîmes
  - Centre Hospitalier Lyon Sud Secteur 1G, Pierre-Bénite
  - Chu Pontchaillou - Service Hematologie, Rennes
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Hôpital Bretonneau, Tours
  - Chru Brabois, Vandœuvre-lès-Nancy
- Germany (5):
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Hämatologisch-Onkologische Praxis Augsburg, Augsburg, Bavaria
  - Universitätsklinikum Halle (Saale), Krukenberg-Krebszentrum Halle (KKH), Halle, Saxony
  - Universitätsklinikum Jena, Klinik für Innere Medizin II, Jena, Thuringia
  - University Hospital Hamburg-Eppendorf, Hamburg
- Greece (3):
  - Laiko General Hospital, Athens
  - UGH of Ioannina, Ioannina
  - University General Hospital of Patras, Rio
- Hong Kong (2):
  - Princess Margaret Hospital, Hong Kong, Kowloon
  - Prince of Wales Hospital, Hong Kong, New Territories
- Hungary (2):
  - : Pecs University, 1st Department of Medicine, Pécs, Pecs
  - Szabolcs Szatmár Bereg Megyei Kórházak és Egyetemi Oktatókórház; Jósa András Oktatókórház, Hematológia, Nyíregyháza
- Israel (9):
  - Soroka Medical Center, Beersheba
  - Shamir Medical Center, Be’er Ya‘aqov
  - Rambam Health Corporation, Haifa
  - Lady Davis Carmel Medical Center, Haifa
  - Wolfson Medical Center, Holon
  - Hadassah University Hospital-Ein Kerem, Jerusalem
  - Shaarei Zedek, Nahariya
  - Rabin Medical Center - Beilinson Campus,, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (15):
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo
  - A.O.U. Policlinico S. Orsola-Malpighi, Bologna
  - Regional Hospital Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliera Universitaria Arcispedale Sant'Anna, Ferrara
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - IRCCS Istituto Romagnolo per lo studio dei tumori "Dino Amadori", Meldola
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera San Gerardo di Monza, Monza
  - University Hospital Maggiore della Carità, Novara
  - AOU S.Luigi Gonzaga, Orbassano
  - University Hospital of Padova, Padua
  - University Hospital 'Paolo Giaccone' Polyclinic, Palermo
  - Ospedale Sant'Eugenio, Rome
  - Hospital Ordine Mauriziano of Turin, Turin
  - Ospedale di Circolo e Fondazione Macchi - ASST Sette Laghi, Varese
- Malaysia (6):
  - Hospital Sultanah Aminah, Johor Bahru, Johor
  - Hospital Sultanah Bahiyah, Alor Star, Kedah
  - Hospital Pulau Pinang, George Town, Pulau Pinang
  - :Hospital Ampang, Ampang, Selangor
  - Sunway Medical Centre, Petaling Jaya, Selangor
  - Hospital Queen Elizabeth, Kota Kinabalu
- Netherlands (2):
  - Amsterdam UMC, Amsterdam
  - Maastricht University Medical Center, Maastricht
- Poland (5):
  - Wojewódzki Szpital Specjalistyczny w Bialej Podlaskiej, Biała Podlaska
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Pratia Onkologia Katowice, Katowice
  - Centrum Medyczne Pratia, Skorzewo
  - Nasz Lekarz Przychodnie Medyczne, Torun
- South Korea (16):
  - Gyeongsang National University Hospital, Jinju, Gyeongsangnam-do
  - Inje University Haeundae Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Inje University Busan Paik Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Daegu Catholic University Medical Center, Daegu
  - The Catholic University Of Korea St. Vincent Hospital, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Jeonbuk National University Hospital, Jeonju
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea, Seoul
  - The Catholic University of South Korea Seoul St. Mary's Hospital, Seoul
  - Ulsan University Hospital, Ulsan
- Spain (12):
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - ICO Badalona - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Clinic de Barcelona, Barcelona
  - Vall d'Hebron Institute of Oncology, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Universitario de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria
  - Quirónsalud Madrid University Hospital, Madrid
  - Morales Meseguer General University Hospital, Murcia
  - Hospital Universitario de Salamanc, Salamanca
  - Hospital Virgen Macarena, Seville
  - University Hospital of Toledo, Toledo
  - Hospital Clínico Universitario de Valencia, Valencia
- Taiwan (4):
  - Chang Gung Memorial Hospital Chiayi, Chiayi City
  - China Medical University Hospital, Chiayi City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- Thailand (5):
  - Songklanagarind Hospital, Songkhla, Hat Yai District
  - Chulabhorn Hospital, Bangkok, Lak Si
  - Srinagarind hospital,Khon Kaen University, Khon Kaen, Mueang Khon Kaen District
  - King Chulalongkorn Memorial Hospital, Bangkok, Pathumwan
  - Rajavithi Hospital, Bangkok, Ratchathewi District
- Turkey (Türkiye) (10):
  - Ankara University Faculty of Medicine Cebeci Research and Application Hospital, Ankara
  - Dr. Abdurrahman Yurtaslan Oncology Health Application and Research Center, Ankara
  - Antalya Medstar Hospital, Antalya
  - Edirne Trakya University Faculty of Medicine Hospital, Edirne
  - Gaziantep University Sahinbey Research and Application Center Hospital, Gaziantep
  - Izmir Ege University Faculty of Medicine Hospital, Izmir
  - Erciyes University Faculty of Medicine Hospital, Kayseri
  - Kocaeli University Application, Kocaeli
  - Mersin University, Mersin
  - Samsun 19 Mayıs University Health Application Research Hospital, Samsun
- United Kingdom (9):
  - Western General Hospital, Edinburgh, Scotland
  - University Hospital of Wales, Cardiff, Wales
  - Pilgrim Hospital, Boston
  - Addenbrooke's Hospital, Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - The Clatterbridge Cancer Centre, Liverpool
  - Guy's & St Thomas NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, Hammersmith Hospital, London
  - University College London Hospitals, London
  - Oxford University Hospitals NHS Foundation Trust, Department of Haematology, Cancer and Haematology Centre, Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Result] Harrison CN, Gupta VK, Gerds AT, Rampal R, Verstovsek S, Talpaz M, Kiladjian JJ, Mesa R, Kuykendall AT, Vannucchi AM, Palandri F, Grosicki S, Devos T, Jourdan E, Wondergem MJ, Al-Ali HK, Buxhofer-Ausch V, Alvarez-Larran A, Patriarca A, Kremyanskaya M, Mead AJ, Akhani S, Sheikine Y, Colak G, Mascarenhas J. Phase III MANIFEST-2: pelabresib + ruxolitinib vs placebo + ruxolitinib in JAK inhibitor treatment-naive myelofibrosis. Future Oncol. 2022 Sep;18(27):2987-2997. doi: 10.2217/fon-2022-0484. Epub 2022 Aug 11. PMID 35950489
- [Result] Rampal RK, Grosicki S, Chraniuk D, Abruzzese E, Bose P, Gerds AT, Vannucchi AM, Palandri F, Lee SE, Gupta V, Lucchesi A, Oh ST, Kuykendall AT, Patriarca A, Alvarez-Larran A, Mesa R, Kiladjian JJ, Talpaz M, Scandura JM, Lavie D, Harris M, Kays SK, Li Q, Boxhammer R, Brown B, Jegg AM, Harrison CN, Mascarenhas J. Pelabresib plus ruxolitinib for JAK inhibitor-naive myelofibrosis: a randomized phase 3 trial. Nat Med. 2025 May;31(5):1531-1538. doi: 10.1038/s41591-025-03572-3. Epub 2025 Mar 10. PMID 40065169

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 135 centers enrolled patients in the study in Australia, Austria, Belgium, Canada, Czech Republic, France, Germany, Greece, Hong Kong, Hungary, Israel, Italy, Malaysia, Netherlands, Poland, South Korea, Spain, Taiwan, Thailand, Turkey, United Kingdom, and United States.
Groups:
- Pelabresib + Ruxolitinib (Experimental Arm): Pelabresib 125 mg orally (PO) once daily (QD) + ruxolitinib 10 or 15 mg orally (PO) twice a day (BID) for 14 consecutive days followed by ruxolitinib 10 or 15 mg orally (PO) twice a day (BID) for 7 days in a 21-day cycle
- Placebo + Ruxolitinib (Control Arm): Matching placebo orally (PO) once daily (QD) + ruxolitinib 10 or 15 mg orally (PO) twice a day (BID) for 14 consecutive days followed by ruxolitinib 10 or 15 mg orally (PO) twice a day (BID) for 7 days in a 21-day cycle
Period: Overall Study
Arm/Group | Pelabresib + Ruxolitinib (Experimental Arm) | Placebo + Ruxolitinib (Control Arm)
Started (Intent-to-Treat (ITT) Analysis Set: all randomized patients, for whom a randomization number has been assigned.) | 214 | 216
Modified Intent-to-Treat (mITT) Analysis Set (All randomized patients who have received at least 1 dose of any study drug(s)) | 212 | 214
Safety Analysis Set (A subset of the ITT population that includes all randomized patients who were administered at least one dose of study drug.) | 212 | 214
Per-Protocol Set (PP Set) | 196 | 194
Pharmacokinetic (PK) Analysis Set (All patients in the Safety Set who received placebo/pelabresib + ruxolitinib treatment and had plasma samples drawn and tested for study drug concentrations.) | 212 | 211
Biomarker Analysis Set (All patients in the Safety Set who received any treatment component and had evaluable biomarker data collected.) | 212 | 214
Ongoing on Double-blind Treatment (Ongoing on double-blind treatment at the time of Primary Completion Date) | 154 | 160
Discontinued Double-blind Treatment (Discontinued double-blind treatment at the time of Primary Completion Date) | 58 | 54
On PFS/OS Follow-up (On Progression-Free Survival (PFS)/Overall Survival (OS) follow-up) | 22 | 30
Completed (Completed Week 24 double-blind treatment) | 181 | 193
Not Completed | 33 | 23

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Population. All randomized patients. This is the primary population for all efficacy endpoints. All analyses using this population will be based on the treatment assigned by the Interactive Response Technology (IRT) system.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pelabresib + Ruxolitinib (Experimental Arm) | Placebo + Ruxolitinib (Control Arm) | Total
Number analyzed (Participants) | 214 | 216 | 430
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 94 | 92 | 186
  >=65 years | 120 | 124 | 244
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (11.84) | 64.8 (11.08) | 64.7 (11.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 94 | 179
  Male | 129 | 122 | 251
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 194 | 199 | 393
  Unknown or Not Reported | 17 | 11 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 35 | 42 | 77
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 160 | 163 | 323
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 16 | 11 | 27
Dynamic International Prognostic Scoring System (DIPSS) risk category [Count of Participants; unit: Participants] — Dynamic International Prognostic Scoring System (DIPSS) is used to predict survival in PMF patients, calculated from five variables: a. Age >65: 1 point b. Leukocyte count >25 × 10^9/L: 1 point c. Hemoglobin <10 g/dL: 2 points d. Circulating blast cells ≥1%: 1 point e. Constitutional symptoms*: 1 point The total DIPSS score categorizes patients into four risk groups, with lower scores indicating better outcomes and longer survival: • 0 points: low risk • 1-2 points: intermediate-1 risk • 3-4 points: intermediate-2 risk • 5-6 points: high risk
  Participants
    Intermediate-1 | 128 | 127 | 255
    Intermediate-2 | 75 | 74 | 149
    High | 11 | 15 | 26
Platelet count [Count of Participants; unit: Participants]
  >200 × 10^9 cells/L | 154 | 157 | 311
  100-200 × 10^9 cells/L | 59 | 57 | 116
  <100 × 10^9 cells/L | 1 | 2 | 3
Hemoglobin [Count of Participants; unit: Participants]
  >10 g/dL | 144 | 140 | 284
  ≤10 g/dL | 70 | 76 | 146
Diagnosis [Count of Participants; unit: Participants]
  Primary Myelofibrosis (PMF) | 107 | 110 | 217
  Post-Polycythemia Vera Myelofibrosis (PPV-MF) | 45 | 53 | 98
  Post-Essential Thrombocythemia Myelofibrosis (PET-MF) | 62 | 53 | 115
Spleen volume from central reads [Mean (Standard Deviation); unit: cm^3] | 1522.43 (950.18) | 1539.28 (920.78) | 1530.90 (934.47)
Baseline Total Symptom Score (TSS) [Mean (Standard Deviation); unit: units on a scale] — Baseline TSS = Averaged daily TSS from the 7-day period prior to randomization (Day -7 to Day -1). Daily TSS is a 24-hour recall format of the MFSAF v4.0, which equals the sum of the 7 individual item responses on the 0-10 scale, with a possible total daily score ranging from 0 to 70. For each individual question, the response scale is 0 (Absent) to 10 (Worst Imaginable).
  units on a scale | 28.26 (12.70) | 27.36 (12.30) | 27.81 (12.50)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Splenic Response by Central Radiology Reads at Week 24
Description: Splenic response was characterized by a reduction of at least 35% in spleen volume from baseline (SVR35), as determined by magnetic resonance imaging (MRI) or computerized tomography (CT), and evaluated through a blinded central radiology review at Week 24.
Time Frame: Week 24
Population: Intent-to-Treat (ITT) Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pelabresib + Ruxolitinib (Experimental Arm) | Placebo + Ruxolitinib (Control Arm)
Number analyzed (Participants) | 214 | 216
Participants | 141 | 76
Statistical Analysis 1: Comparison: Pelabresib + Ruxolitinib (Experimental Arm) vs Placebo + Ruxolitinib (Control Arm); Splenic Response Rate at Week 24; Test type: Other — The response rate between the 2 treatment groups was compared using CMH test; p < 0.001, Cochran-Mantel-Haenszel; CMH 95% CI adjusted by strata; Mehrotra-Railkar test used if Breslow-Day significant; DIPSS High merged with Int-2 due to low counts; Difference in proportion = 30.4, 95% CI 2-sided [21.6 to 39.3] — The proportion difference = experimental group (Pela + RUX) - control group (placebo + RUX)

2. Secondary Outcome: Key Secondary: Absolute Change From Baseline in Total Symptom Score (TSS) at Week 24
Description: The Total Symptom Score (TSS) at Week 24, compared to baseline, was measured using the Myelofibrosis Symptom Assessment Form v4.0. This score represented the sum of seven individual symptom items, each rated on a 0-10 scale, resulting in a possible total daily score ranging from 0 to 70. A higher TSS reflected a greater disease burden and therefore a worse outcome. The baseline TSS was calculated as the average of non-missing daily total symptom scores over the seven-day period preceding the day of randomization. The TSS for each treatment week was determined as the average of non-missing daily total symptom scores for that week. However, if fewer than four daily scores were available for a given week, the weekly TSS was considered missing.
Time Frame: Baseline, Week 24
Population: Intent-to-Treat (ITT) Analysis Set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pelabresib + Ruxolitinib (Experimental Arm) | Placebo + Ruxolitinib (Control Arm)
Number analyzed (Participants) | 214 | 216
score on a scale | -15.99 (1.028) | -14.05 (0.986)
Statistical Analysis 1: Comparison: Pelabresib + Ruxolitinib (Experimental Arm) vs Placebo + Ruxolitinib (Control Arm); Absolute Change from Baseline in Total Symptom Score (TSS) at Week 24; Test type: Other; p = 0.0545, ANCOVA; LS Mean Difference = -1.94, 95% CI 2-sided [-3.92 to 0.04], Standard Error of Mean 1.009

3. Secondary Outcome: Key Secondary: Number of Participants With TSS50 Response at Week 24
Description: The probability of a TSS response at Week 24 was estimated by calculating the TSS response rate, defined as the percentage of patients who achieved a TSS50 response at Week 24 in each of the two treatment groups. The Total Symptom Score (TSS) response was defined as a ≥50% reduction from baseline in TSS, as measured by the Myelofibrosis Symptom Assessment Form v4.0.
Time Frame: Week 24
Population: Intent-to-Treat (ITT) Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pelabresib + Ruxolitinib (Experimental Arm) | Placebo + Ruxolitinib (Control Arm)
Number analyzed (Participants) | 214 | 216
Participants | 112 | 100
Statistical Analysis 1: Comparison: Pelabresib + Ruxolitinib (Experimental Arm) vs Placebo + Ruxolitinib (Control Arm); Percentage of TSS50 at Week 24; Test type: Other — The response rate between the 2 treatment groups was compared using CMH test; p = 0.216, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 6.0, 95% CI 2-sided [-3.4 to 15.5] — Proportion Difference = Experimental Group (Pela + RUX) - Control Group (placebo + RUX)

4. Secondary Outcome: Percent Change From Baseline in Total Symptom Score (TSS) at Week 24
Description: Percent Change From Baseline in Total Symptom Score (TSS) at Week 24 measured the change in a patient's symptoms after 24 weeks of treatment, relative to baseline. A negative value indicates symptom improvement, and a reduction of ≥50% is typically considered a meaningful clinical response.
Time Frame: Baseline, Week 24
Population: Intent-to-Treat (ITT) Analysis Set
Measure: Mean (95% Confidence Interval); unit: Percent change from baseline to Week 24
Arm/Group | Pelabresib + Ruxolitinib (Experimental Arm) | Placebo + Ruxolitinib (Control Arm)
Number analyzed (Participants) | 184 | 193
Percent change from baseline to Week 24 | -50.3 [-56.6 to -44.0] | -45.9 [-51.8 to -40.0]

5. Secondary Outcome: Number of Participants With Improvement From Baseline in Bone Marrow Fibrosis of at Least 1 Grade at Week 24
Description: Improvement in bone marrow fibrosis by at least 1 grade, as assessed by central read compared to baseline, was analyzed by treatment group and overall. The improvement in bone marrow fibrosis grade was defined as a decrease by at least 1 grade in bone marrow fibrosis grade when compared to baseline, where a grade of MF-3 was the most severe, and MF-0 was the least severe.
Time Frame: Baseline, Week 24
Population: Intent-to-Treat (ITT) Analysis Set: Only participants with available data at the specified time point were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Pelabresib + Ruxolitinib (Experimental Arm) | Placebo + Ruxolitinib (Control Arm)
Number analyzed (Participants) | 192 | 188
Participants | 36 | 21
Statistical Analysis 1: Comparison: Pelabresib + Ruxolitinib (Experimental Arm) vs Placebo + Ruxolitinib (Control Arm); ≥1 Grade improvement From Baseline in Bone Marrow Fibrosis at Week 24; Test type: Other; p = 0.037, Cochran-Mantel-Haenszel; CMH 95% CI adjusted across the strata including baseline DIPSS, platelet count, and spleen volume; Difference in proportions = 7.63, 95% CI 2-sided [0.52 to 14.73] — Proportion Difference = Experimental Group (Pela + RUX) - Control Group (placebo + RUX)

6. Secondary Outcome: Number of Participants With Splenic Response by Central Radiology Reads at Week 48
Description: Splenic response is characterized by a reduction of at least 35% in spleen volume from baseline (SVR35), as determined by magnetic resonance imaging (MRI) or computerized tomography (CT), and evaluated through a blinded central radiology review at Week 48.
Time Frame: Week 48
Reporting Status: Not Posted, anticipated posting 2027-12

7. Secondary Outcome: Number of Participants With TSS50 Response at Week 48
Description: The probability of a TSS response at Week 48 is estimated by calculating the TSS response rate, defined as the percentage of patients who achieve a TSS50 response at Week 48 in each of the two treatment groups. The Total Symptom Score (TSS) response is defined as a ≥50% reduction from baseline in TSS, as measured by the Myelofibrosis Symptom Assessment Form v4.0.
Time Frame: Week 48
Reporting Status: Not Posted, anticipated posting 2027-12

8. Secondary Outcome: Absolute Change From Baseline in Total Symptom Score (TSS) at Week 48
Description: The Total Symptom Score (TSS) at Week 48, compared to baseline, is measured using the Myelofibrosis Symptom Assessment Form v4.0. This score represents the sum of seven individual symptom items, each rated on a 0-10 scale, resulting in a possible total daily score ranging from 0 to 70. A higher TSS reflects a greater disease burden and therefore a worse outcome. The baseline TSS is calculated as the average of non-missing daily total symptom scores over the seven-day period preceding the day of randomization. The TSS for each treatment week is determined as the average of non-missing daily total symptom scores for that week. However, if fewer than four daily scores are available for a given week, the weekly TSS is considered missing.
Time Frame: Baseline, Week 48
Reporting Status: Not Posted, anticipated posting 2027-12

9. Secondary Outcome: Rate of Red Blood Cell (RBC) Transfusion Over First 24 Weeks of Treatment
Description: The rate of RBC transfusions was defined as the average number of RBC units transfused per patient month (4 weeks) during the first 24 weeks of treatment. The average number of RBC units per patient-month was calculated by dividing the total (ie, for all patients) number of RBC units in the whole exposure time by the sum of patient-months.
Time Frame: Week 24
Population: Intent-to-Treat (ITT) Analysis Set
Measure: Number (95% Confidence Interval); unit: RBC units transfused/patient-months
Arm/Group | Pelabresib + Ruxolitinib (Experimental Arm) | Placebo + Ruxolitinib (Control Arm)
Number analyzed (Participants) | 195 | 201
RBC units transfused/patient-months | 1.359 [0.982 to 1.736] | 1.014 [0.840 to 1.188]

10. Secondary Outcome: Number of Participants Who Transitioned From Red Blood Cell (RBC) Transfusion Dependence to Transfusion Independence
Description: Transfusion dependence (TD) was defined as having received ≥6 units of RBCs during the 12-week baseline period prior to dosing and Transfusion independence (TI) was defined as the absence of RBC transfusions during any continuous 12-week period of the double-blind treatment phase.
  The conversion from TD to TI was evaluated and defined as the proportion of patients who transitioned from transfusion dependence to transfusion independence. Patients who remained in the double-blind treatment period and had not received any RBC transfusions during the most recent 12 weeks were considered responders. Patients who discontinued from the double-blind treatment before Week 12 were classified as non-responders.
Time Frame: From 12-week baseline period prior to dosing to any 12-week period post baseline, up to 24 weeks
Population: Intent-to-Treat (ITT) Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pelabresib + Ruxolitinib (Experimental Arm) | Placebo + Ruxolitinib (Control Arm)
Number analyzed (Participants) | 214 | 216
Participants | 0 | 0

11. Secondary Outcome: Category Change From Baseline of Patient Global Impression of Change (PGIC) at Week 24
Description: The Patient Global Impression of Change (PGIC) was a single-item measure of the patient's perceived change in MF symptoms since starting treatment. Patients responded to: "Since beginning this study treatment, your myelofibrosis symptoms were: (1) Very much improved, (2) Much improved, (3) Minimally improved, (4) No change, (5) Minimally worse, (6) Much worse, (7) Very much worse."
Time Frame: Baseline, Week 24
Population: Intent-to-Treat (ITT) Analysis Set - Only participants with evaluable data at the pre-specified time points
Measure: Count of Participants; unit: Participants
Arm/Group | Pelabresib + Ruxolitinib (Experimental Arm) | Placebo + Ruxolitinib (Control Arm)
Number analyzed (Participants) | 177 | 194
Participants
  Very much improved | 24 | 26
  Much improved | 63 | 62
  Minimally improved | 63 | 79
  No change | 14 | 13
  Minimally worse | 7 | 14
  Much worse | 5 | 0
  Very much worse | 1 | 0

12. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-Free Survival (PFS), defined as the time from randomization until documented progression, or until death from any cause for patients without documented progression
Time Frame: Through study completion, an average of 6 years
Reporting Status: Not Posted, anticipated posting 2027-12

13. Secondary Outcome: Overall Survival (OS)
Description: OS, defined as the time from randomization until death from any cause
Time Frame: Through study completion, an average of 6 years
Reporting Status: Not Posted, anticipated posting 2027-12

14. Secondary Outcome: Proportion of Patients With Transformation to Blast Phase (AML)
Description: Patients are categorized as having transformed to Acute Myelogenous Leukemia (AML) when the peripheral blood blast percentage increases to ≥20% and this elevation persists for at least two weeks, or when leukemic transformation is confirmed through disease status assessment.
Time Frame: Through study completion, an average of 6 years
Reporting Status: Not Posted, anticipated posting 2027-12

15. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: A treatment-emergent adverse event (TEAE) for the double-blind treatment period is defined as an AE that has a start date on or after the first dose of the pelabresib/placebo and before 30 days after the last dose of pelabresib/placebo or before the start of alternative (off-study) treatment for MF, whichever occurs first. If the AE has a start date before the date of first dose but increases in severity after first dose and before 30 days post last dose will be considered a TEAE as well. An AE that occurs after the administration of the first dose of open-label pelabresib treatment will be considered treatment-emergent for the crossover treatment period. However, a TEAE for the crossover treatment period that occurs within 30 days after the last dose of pelabresib/placebo will be considered treatment emergent for the double-blind treatment period as well.
Time Frame: Through study completion, an average of 6 years
Reporting Status: Not Posted, anticipated posting 2027-12

16. Secondary Outcome: Pharmacokinetic (PK) Parameters for Pelabresib: Area Under the Plasma Concentration-time Curve From Time Zero to Time t (AUC0-t)
Description: Pharmacokinetic (PK) parameters will be calculated based on Pelabresib plasma concentrations and actual sampling time points.
  AUC0-t will be listed and summarized using descriptive statistics.
Time Frame: Cycle 1 Day 1, Cycle 1 Day 14 and Cycle 9 Day 1: Predose, 30 minutes to 1 hour post-dose, 3 to 4.5 hours post-dose. Cycle 3 and Cycle 7 Day 1: Predose, 5 minutes post ECG assessment. 1 Cycle = 21 days
Reporting Status: Not Posted, anticipated posting 2027-12

17. Secondary Outcome: Pharmacokinetic (PK) Parameters for Pelabresib: Time to Reach Maximum (Peak) Plasma Concentration Following Drug Administration (Tmax)
Description: Pharmacokinetic (PK) parameters will be calculated based on Pelabresib plasma concentrations and actual sampling time points.
  AUC0-t will be listed and summarized using descriptive statistics. Tmax will be listed and summarized using descriptive statistics.
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2027-12

18. Secondary Outcome: Pharmacokinetic (PK) Parameters for Pelabresib: Maximum (Peak) Plasma Drug Concentration (Cmax)
Description: Pharmacokinetic (PK) parameters will be calculated based on Pelabresib plasma concentrations and actual sampling time points.
  AUC0-t will be listed and summarized using descriptive statistics. Cmax will be listed and summarized using descriptive statistics.
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2027-12

19. Secondary Outcome: Pharmacokinetic (PK) Parameters for Pelabresib: Effective Half-Life (T1/2)
Description: Pharmacokinetic (PK) parameters will be calculated based on Pelabresib plasma concentrations and actual sampling time points.
  T1/2 will be listed and summarized using descriptive statistics.
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2027-12

20. Secondary Outcome: Pharmacokinetic (PK) Parameters for Pelabresib: Apparent Volume of Distribution After Non-intravenous Administration (Vd/F)
Description: Pharmacokinetic (PK) parameters will be calculated based on Pelabresib plasma concentrations and actual sampling time points.
  Vd/F will be listed and summarized using descriptive statistics.
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2027-12

21. Secondary Outcome: Pharmacokinetic (PK) Parameters for Pelabresib: Apparent Total Clearance of the Drug From Plasma After Oral Administration (CL/F)
Description: Pharmacokinetic (PK) parameters will be calculated based on Pelabresib plasma concentrations and actual sampling time points.
  CL/F will be listed and summarized using descriptive statistics.
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2027-12

22. Secondary Outcome: Ruxolitinib Plasma Concentrations in the Presence or Absence of Pelabresib
Description: Blood samples (approximately 4 mL each) will be collected at the time points specified in the Schedule of Assessments (SOA) to determine plasma concentrations of Ruxolitinib plasma concentrations in the presence or absence of Pelabresib
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2027-12

23. Secondary Outcome: Duration of the Splenic Response
Description: Duration of splenic response, defined as the time from onset of splenic response until the time at which the patient has a <35% decrease from baseline in spleen volume and a >25% increase from nadir, as confirmed by the central review) or death, whichever comes first
Time Frame: Through study completion, an average of 6 years
Reporting Status: Not Posted, anticipated posting 2027-12

24. Secondary Outcome: Number of Participants With Modified Total Symptom Score (mTSS) Response at Week 24
Description: The modified TSS (mTSS) was defined as TSS without the fatigue sub-domain and with a total scale of 60 points versus 70 points for TSS. Patients were classified as responders if the percentage of change from baseline in mTSS was ≤ -50% at Week 24.
Time Frame: Week 24
Population: Intent-to-Treat (ITT) Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pelabresib + Ruxolitinib (Experimental Arm) | Placebo + Ruxolitinib (Control Arm)
Number analyzed (Participants) | 214 | 216
Participants | 120 | 104
Statistical Analysis 1: Comparison: Pelabresib + Ruxolitinib (Experimental Arm) vs Placebo + Ruxolitinib (Control Arm); Modified Total Symptom Score (mTSS) Response at Week 24; Test type: Other; p = 0.107, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in Proportions = 7.8, 95% CI 2-sided [-1.7 to 17.2] — The proportion difference = experimental group (Pela + RUX) - control group (placebo + RUX). Wald 95% CIs were applied

25. Secondary Outcome: Duration of the TSS50 Response
Description: Duration of TSS response, defined as the time from onset of TSS50 response until the time at which the patient has a <50% reduction in TSS from baseline and an increase of ≥25% from nadir
Time Frame: Through study completion, an average of 6 years
Reporting Status: Not Posted, anticipated posting 2027-12

ADVERSE EVENTS:
Time Frame: From first dose of study treatment up to the cut-off date for the interim analysis (31-Aug-2023), approximately 28 months
Description: Adverse Events were reported that had a start date on or after the first dose of the pelabresib/placebo and before 30 days after the last dose of pelabresib/placebo or before the start of alternative (off study) treatment for MF, whichever occured first. In addition, Serious Adverse Events, including deaths, that were reported at any time after 30 days after the last dose of pelabresib/placebo are presented.
Arm/Group | Pelabresib + Ruxolitinib (Experimental Arm) | Placebo + Ruxolitinib (Control Arm)
All-Cause Mortality (participants affected / at risk) | 11/212 | 10/214
Serious Adverse Events (participants affected / at risk) | 63/212 | 63/214
Other Adverse Events (participants affected / at risk) | 201/212 | 204/214
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pelabresib + Ruxolitinib (Experimental Arm) (N=212) | Placebo + Ruxolitinib (Control Arm) (N=214)
Anaemia (Blood and lymphatic system disorders) | 5 | 5
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 0 | 3
Arrhythmia (Cardiac disorders) | 2 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 2
Cardiac Arrest (Cardiac disorders) | 2 | 0
Cardiac Failure Congestive (Cardiac disorders) | 2 | 0
Myocardial Infarction (Cardiac disorders) | 2 | 0
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0
Left Ventricular Failure (Cardiac disorders) | 0 | 1
Myocardial Ischaemia (Cardiac disorders) | 1 | 0
Sinus Node Dysfunction (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Thyroid Mass (Endocrine disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0
Chronic Gastritis (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastric Ulcer (Gastrointestinal disorders) | 0 | 1
Gastric Varices Haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophageal Varices Haemorrhage (Gastrointestinal disorders) | 0 | 1
Varices Oesophageal (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 1
Chest Pain (General disorders) | 0 | 1
Drug Withdrawal Syndrome (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Sudden Cardiac Death (General disorders) | 0 | 1
Bile Duct Stone (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 0
Pneumonia (Infections and infestations) | 7 | 6
Sepsis (Infections and infestations) | 3 | 2
Herpes Zoster (Infections and infestations) | 4 | 0
Covid-19 (Infections and infestations) | 0 | 3
Covid-19 Pneumonia (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 0 | 2
Urinary Tract Infection (Infections and infestations) | 0 | 2
Abscess Neck (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Campylobacter Infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Enterococcal Infection (Infections and infestations) | 0 | 1
Fungal Infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 1
Gastrointestinal Viral Infection (Infections and infestations) | 0 | 1
Herpes Zoster Meningoencephalitis (Infections and infestations) | 0 | 1
Herpes Zoster Oticus (Infections and infestations) | 1 | 0
Liver Abscess (Infections and infestations) | 0 | 1
Norovirus Infection (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 1 | 0
Pneumonia Bacterial (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Pyelonephritis Acute (Infections and infestations) | 1 | 0
Septic Shock (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Accidental Overdose (Injury, poisoning and procedural complications) | 2 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 1
Skin Graft Necrosis (Injury, poisoning and procedural complications) | 0 | 1
Splenic Rupture (Injury, poisoning and procedural complications) | 0 | 1
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0
Platelet Count Decreased (Investigations) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Haematoma Muscle (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adenocarcinoma Gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Atypical Fibroxanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bowen's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant Fibrous Histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Precursor T-Lymphoblastic Lymphoma/Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous Cell Carcinoma Of The Tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Syncope (Nervous system disorders) | 2 | 2
Cerebrovascular Accident (Nervous system disorders) | 1 | 0
Haemorrhage Intracranial (Nervous system disorders) | 1 | 0
Post Herpetic Neuralgia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 2 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Embolism Arterial (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Shock Haemorrhagic (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pelabresib + Ruxolitinib (Experimental Arm) (N=212) | Placebo + Ruxolitinib (Control Arm) (N=214)
Anaemia (Blood and lymphatic system disorders) | 90 | 116
Thrombocytopenia (Blood and lymphatic system disorders) | 68 | 50
Constipation (Gastrointestinal disorders) | 39 | 52
Diarrhoea (Gastrointestinal disorders) | 49 | 39
Nausea (Gastrointestinal disorders) | 30 | 32
Abdominal Pain Upper (Gastrointestinal disorders) | 17 | 14
Vomiting (Gastrointestinal disorders) | 15 | 16
Abdominal Pain (Gastrointestinal disorders) | 8 | 19
Fatigue (General disorders) | 25 | 34
Asthenia (General disorders) | 25 | 30
Pyrexia (General disorders) | 16 | 19
Oedema Peripheral (General disorders) | 12 | 16
Covid-19 (Infections and infestations) | 24 | 32
Upper Respiratory Tract Infection (Infections and infestations) | 18 | 15
Herpes Zoster (Infections and infestations) | 16 | 11
Urinary Tract Infection (Infections and infestations) | 13 | 14
Contusion (Injury, poisoning and procedural complications) | 14 | 15
Platelet Count Decreased (Investigations) | 44 | 34
Alanine Aminotransferase Increased (Investigations) | 20 | 19
Weight Increased (Investigations) | 13 | 20
Aspartate Aminotransferase Increased (Investigations) | 15 | 15
Blood Creatinine Increased (Investigations) | 9 | 17
Decreased Appetite (Metabolism and nutrition disorders) | 16 | 11
Hyperkalaemia (Metabolism and nutrition disorders) | 8 | 17
Hyperuricaemia (Metabolism and nutrition disorders) | 9 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 24
Back Pain (Musculoskeletal and connective tissue disorders) | 18 | 20
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 11 | 15
Dysgeusia (Nervous system disorders) | 39 | 8
Headache (Nervous system disorders) | 24 | 23
Dizziness (Nervous system disorders) | 24 | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 27 | 24
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 27
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 21
Rash (Skin and subcutaneous tissue disorders) | 15 | 7
Hypertension (Vascular disorders) | 16 | 11
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 24 | 9
Bone Pain (Musculoskeletal and connective tissue disorders) | 10 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-10-04): https://cdn.clinicaltrials.gov/large-docs/95/NCT04603495/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-26): https://cdn.clinicaltrials.gov/large-docs/95/NCT04603495/SAP_001.pdf